CLINICAL TRIAL: NCT06603480
Title: Effects of Exercise and Metformin on Methylglyoxal Levels in Prediabetic Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MEGS
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Methylglyoxal; PreDiabetes; Exercise; Metformin
Keywords: Physical activity; PreDiabetes; Metformin; Methylglyoxal
MeSH Terms: conditions — Prediabetic State; Motor Activity | interventions — Exercise; Metformin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aerobic Exercise (Active Comparator): 12 week aerobic exercise
  Interventions: Behavioral: Exercise
- Metformin (Experimental): Metformin 2*1 given
  Interventions: Other: Metformin
- Control (No Intervention): Only routine

INTERVENTIONS:
Behavioral: Exercise — Aerobic exercise (moderate intensity) at 50-70% of maximum heart rate for 60 minutes, 3 days a week for 12 weeks
  Arms: Aerobic Exercise
Other: Metformin — Patients who started Metformin 2*1
  Arms: Metformin

SUMMARY:
The aim of this study is to compare the effects of exercise, standard lifestyle changes and metformin on MGO in prediabetic individuals.

DETAILED DESCRIPTION:
There is no comparative study in the literature evaluating the effects of exercise and metformin on MGO in prediabetic patients. The aim of this study is to compare the effects of exercise, standard lifestyle changes and metformin on MGO in prediabetic individuals.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were newly diagnosed with prediabetes by Oral Glucose Tolerance Test (OGTT) and/or HbA1C,
* who were assessed as physically inactive (Level 1) according to the International Physical Activity Questionnaire
* who had sufficient motivation to participate in the exercise program (assessed by one-on-one interviews conducted by the researchers),
* who were deemed suitable to participate in the exercise program after a cardiac examination by a cardiologist (with resting electrocardiogram and questioning of cardiac symptoms, and advanced tests such as exercise electrocardiogram test when necessary),
* who had the same weight (±2.5 kg) for 6 months before participating in the study.

Exclusion Criteria:

* having a serious medical condition that would prevent the person from participating in the exercise study (e.g. advanced malignancy or major neurological, psychiatric or endocrine disease, respiratory failure, etc.),
* having used metformin for 6 months before the study, having cardiovascular disease,
* heart failure, cancer, having a BMI <19 kg/m2, receiving hormone replacement therapy,
* having a life expectancy of less than 1 year, being HIV positive, substance use,
* functional dependence, having an orthopedic disease that prevents physical activity,
* having cognitive impairment and other diseases that would affect the study results (respiratory diseases, muscle diseases, non-alcoholic fatty liver disease, etc.),
* using medications or supplements that would affect the study results.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
MGO | 1 week
  Methylgloxal level

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan 2. Abdülhamid Han Training and Research Hospital, Üsküdar, Istanbul, Turkey (Türkiye)